CLINICAL TRIAL: NCT02240433
Title: A Phase 1b Study of LY2157299 in Combination With Sorafenib in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Study of LY2157299 in Participants With Unresectable Hepatocellular Cancer (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14856; H9H-JE-JBAP (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — LY-2157299; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY2157299 + Sorafenib (Experimental): LY2157299 will be administered orally twice daily for 14 days, followed by 14 days with no study drug per 28-day cycle. Sorafenib will be administered orally twice daily for 28 days, in each cycle.
  Interventions: Drug: LY2157299; Drug: Sorafenib

INTERVENTIONS:
Drug: LY2157299 — LY2157299 administered orally
Drug: Sorafenib — Sorafenib administered orally

SUMMARY:
The main purpose of this study is to evaluate safety and tolerability of LY2157299 when combined with sorafenib in Japanese hepatocellular carcinoma (HCC) participants.

ELIGIBILITY:
Inclusion Criteria:

* Have histological evidence of a diagnosis of HCC (except HCC with fibrolamellar or mixed histology) not amenable to curative surgery.
* Have Child-Pugh Class A.
* Have the presence of measurable or evaluable lesion as defined by the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. A measurable or evaluable lesion showing demonstrable progression after locoregional therapy could be also included.
* Have not received sorafenib prior to enrollment.
* Have resolution to Grade less than or equal 1 by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 of all clinically significant toxic effects of prior locoregional therapy, surgery, chemoembolization, systemic chemotherapy.
* Have a performance status of less than or equal 1 on the Eastern Cooperative Oncology Group (ECOG) scale.

Exclusion Criteria:

* Are currently enrolled, or discontinued within 28 days prior to enrollment from, a clinical trial involving an investigational product or nonapproved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have undergone major surgery within 28 days prior to enrollment.
* Have undergone hepatic locoregional therapy (including radiation, surgery, hepatic arterial embolization, chemoembolization, radiofrequency ablation, cryoablation, percutaneous ethanol injection, or percutaneous microwave coagulation therapy) within 28 days prior to enrollment.
* Have moderate or severe cardiac disease.

  * Myocardial infarction within 6 months prior to enrollment, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension.
  * Documented major electrocardiogram (ECG) abnormalities at the investigator's discretion within 28 days prior to enrollment.
  * Major abnormalities documented by echocardiography with Doppler at investigator's direction within 28 days prior to enrollment.
  * Have persistently elevated brain natriuretic peptide (BNP) or elevated troponin I within 14 days prior to enrollment.
  * Predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress.
  * Have a history of cardiac or aortic surgery.
* Have undergone liver transplant.
* Are pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with LY2157299 Dose-Limiting Toxicities (DLT) | Cycle 1 (28 days)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Plasma Concentration-time Curve (AUC) of LY2157299 | Cycle 1 Day1: predose through 6 hours post dose; Cycle1 Day14: predose through 24 hours post dose
PK: Maximum Observed Plasma Concentration (Cmax) of LY2157299 | Cycle 1 Day 1: Predose through 6 hours post dose; Cycle 1 Day 14: Predose through 24 hours post dose
Time to Progression (TTP) | Baseline to objective progressive disease (estimated as 6 months)
Progression-free Survival (PFS) | Baseline to objective progressive disease or death (estimated as 6 months)
The Number of Participants with Best Response of Partial Response (PR), Complete Response (CR), Stable Disease (SD), or Progressive Disease (PD) | Baseline to objective progressive disease (estimated as 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suita-shi